CLINICAL TRIAL: NCT05335993
Title: Phase 2, Single Arm Clinical Trial to Evaluate the Safety and Activity of Oregovomab and Niraparib as a Combinatorial Immune Priming Strategy in Subjects With Platinum Sensitive Recurrent Ovarian Cancer
Brief Title: A Clinical Study Evaluating a Combination of Oregovomab and Niraparib in Adult Women With Platinum Sensitive Recurrent Ovarian Cancer.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CanariaBio Inc. (Industry)
Collaborators: Veristat, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QPT-ORE-004
Record Dates: First submitted 2022-02-10; First posted 2022-04-20 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Ovarian Cancer; Recurrent Epithelial Cancer of Ovary; Recurrent Epithelial Ovarian Cancer; Recurrent Fallopian Tube Cancer; Peritoneal Cancer; Recurrent Carcinoma of Ovary; Adenocarcinoma of Ovary
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — oregovomab; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination of Oregovomab and Niraparib (Experimental): * Niraparib (300/200 mg) will be administered orally once daily.
  * Oregovomab (2 mg) will be administered via IV infusion on Day 1 of Week 1, Week 4, Week 7, Week 12, and Week 20.
  Interventions: Biological: Oregovomab; Drug: Niraparib

INTERVENTIONS:
Biological: Oregovomab — 2 mg, added to 50 mL of Sodium Chloride infused over 20 ± 5 minutes.
  Other Names: MAb-B43.13; Monoclonal antibody B43.13
Drug: Niraparib — 300mg administered orally once daily starting at the first day of treatment (Day 1 Week 1) to the end of Week 12. Subjects whose baseline weight is <77 kg or platelet count is <150,000 μL, the daily dosing will be 200mg.
  Other Names: Zejula

SUMMARY:
Study to evaluate the safety and activity of oregovomab and niraparib as a combinatorial immune priming strategy in subjects with platinum sensitive recurrent ovarian cancer.

DETAILED DESCRIPTION:
Phase 2 single arm open label study to evaluate the combination of oregovomab and niraparib as a combinatorial immune priming strategy in subjects with platinum sensitive recurrent ovarian cancer. Approximately 15 subjects will be screened to enroll approximately 10 evaluable subjects.

The study will include:

* Screening period up to 28 days prior to start of study treatment.
* Treatment period up to 24 weeks.
* Post-treatment follow-up period:
* Safety Follow-up: all subjects will be followed at least 30 days after end of treatment for safety.
* Long Term Follow-up: all subjects will be followed for survival approximately every 3 months for 1 year, until death, withdrawal of consent, lost to follow-up, or sponsor decision to close the study; or whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with CA125-associated recurrent epithelial adenocarcinoma of ovarian, fallopian tube or peritoneal origin.
2. Subjects must have histologically diagnosed high-grade (Grade 2 or 3) serous epithelial ovarian, fallopian tube, or primary peritoneal cancer with recurrent disease and must have been previously treated with chemotherapy and experienced a response lasting at least 6 months to first-line platinum-based therapy.
3. Previously treated disease with up to 3 prior lines of therapy, including at least one platinum-based therapy. Each line of therapy should have been changed due to recurrence, progression, or toxicity. Maintenance therapy with bevacizumab, hormonal therapies and / or a PARP inhibitor is not considered a line of therapy.
4. Must have received prior platinum-based chemotherapy for first line ovarian cancer, however they must have been platinum sensitive for ≥6 months after the most recent platinum-containing regimen prior to the start of study treatment.
5. Must have medical assessment consistent with prognosis for an expected survival of at least 6 months and be clinically appropriate to receive a 12-week hiatus from any cytotoxic treatment according to the best clinical judgement of the treating Investigator.
6. Must have had an elevated serum CA125 >50 units / mL measured at screening within 28 days of start of study treatment.
7. Must have measurable disease, including identification of marker lesions, by radiographic or physical criteria suitable for evaluation according to RECIST v1.1 for documentation of disease response or progression.
8. Must have an ECOG Performance Status of 0, 1 or 2.
9. Must have adequate organ function defined as:

   1. Absolute neutrophil count ≥1,500 / μL
   2. Platelets ≥100,000 / μL
   3. Hemoglobin ≥9 g / dL
   4. Total bilirubin ≤1.5 x ULN (≤2.0 x ULN in subjects with known Gilberts syndrome) OR direct bilirubin ≤1 x ULN
   5. LDH, SGOT and SGPT<2.5 x ULN
   6. Albumin >3.5 g / dL
   7. Serum Creatinine < 1.5 mg/dL
10. For women of childbearing potential, a negative pregnancy test and willingness to avoid pregnancy by using a highly effective method of contraception from the first dose of study treatment to 6 months after last dose of study treatment.
11. Able to take oral medications.
12. Sign informed consent and authorization permitting release of personal health information.

Exclusion Criteria:

1. Subject must not be simultaneously treated in any interventional clinical trial.
2. Subject must not have had major surgery ≤3 weeks prior to initiating protocol therapy and subject must have recovered from any surgical effects.
3. Subject must not have received investigational therapy ≤4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior to initiating protocol therapy.
4. Subject has had radiation therapy encompassing >20% of the bone marrow within 2 weeks;
5. Subject must not have received a transfusion (platelets or red blood cells) ≤2 weeks prior to first dose of study treatment.
6. Subject must not have received colony-stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 4 weeks prior to initiating protocol therapy.
7. Subject has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted >4 weeks and was related to the most recent treatment.
8. Subject must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection or active infection causing fever. Examples include, but are not limited to, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent. Subjects with chronic diseases that are well controlled (e.g., diabetes mellitus, hypertension [<140 sBP and <90 dBP]) are eligible.
9. Evidence of clinically significant cardiovascular and respiratory conditions including myocardial infarction within 1 year, uncontrolled or unstable angina, congestive heart failure (New York Heart Association Class III or IV), arrhythmia (Grade 2 or higher), chronic obstructive pulmonary disease, persistent asthma, or a history of asthma within 5 years.
10. Subject must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
11. Diagnosed or treated for another malignancy within 5 years before the first dose, or previously diagnosed with another malignancy and have any evidence of residual disease. Subjects with non-melanoma skin cancer or cervix carcinoma in situ are not excluded if they have undergone complete resection.
12. Subject must not have known, symptomatic brain or leptomeningeal metastases.
13. Have an active autoimmune disease (e.g., rheumatoid arthritis, SLE, ulcerative colitis, Crohn's Disease, MS, ankylosing spondylitis, thyroiditis) requiring continuing immune suppressive therapy.
14. Recognized immunodeficiency condition including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; subjects who have hereditary, or congenital immunodeficiency's (HIV infection, see below).
15. Chronically treated with systemic doses of immunosuppressive drugs such as cyclosporine, methotrexate, adrenocorticotropic hormone (ACTH) or immune suppressive monoclonal antibodies.
16. Chronic therapeutic corticosteroid use, defined as >5 days of prednisone or equivalent, with the exception of inhalers or those on a pre-planned steroid taper. (Note: Premedication with corticosteroids per institutional standard of care is allowed).
17. Any previous treatments with oregovomab.
18. Known allergy to murine proteins or hypersensitivity to oregovomab, niraparib, or any of the excipients of oregovomab or niraparib.
19. Have contraindications to the use of pressor agents (e.g., SC epinephrine), notably monoamine oxidase inhibitor (MAOI) use.
20. Any of the following conditions (on-study testing is not required):

    1. Known HIV-infected subjects unless on effective anti-retroviral therapy with an undetectable viral load within 6 months, or
    2. Known or suspected hepatitis B if active infection (subjects with chronic hepatitis B infection must have an undetectable HBV viral load on suppressive therapy, if indicated; positive surface antibody alone is not an exclusion), or
    3. Known or suspected hepatitis C infection which has not been treated and cured unless currently on treatment with an undetectable viral load).
21. Unable understand, and / or unwilling to sign a written consent form which must be obtained prior to treatment.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women 18 years of age and older.
Enrollment: 10 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Disease Control Rate (DCR) | At 12 weeks
  To evaluate anti-tumor activity of oregovomab added to niraparib by Disease Control Rate, defined as the portion of subjects with complete response (CR), partial response (PR) and stable disease (SD) at week 12. The DCR will be determined as defined by RECIST 1.1
Assessment of Disease Control Rate (DCR) | At 24 weeks
  To evaluate anti-tumor activity of oregovomab added to niraparib by Disease Control Rate, defined as the portion of subjects with complete response (CR), partial response (PR) and stable disease (SD) at week 24. The DCR will be determined as defined by RECIST 1.1

SECONDARY OUTCOMES:
To Establish the Preliminary Safety and Tolerability of Oregovomab When Added to Niraparib. | Up to 30 days post last End of Treatment
  Frequency of adverse events (AEs), serious adverse events (SAEs), deaths and AEs leading to discontinuation of treatment as defined by CTCAE version 5.0.
To Establish the Preliminary Safety and Tolerability of Oregovomab When Added to Niraparib. | Up to week 24
  A. Change in baseline from week 1 to week 24 the frequency of vital signs taken.
To Establish the Preliminary Safety and Tolerability of Oregovomab When Added to Niraparib. | Up to week 24
  Change in baseline from week 1 to week 24 the severity of vital sign measurements.
To Establish the Preliminary Safety and Tolerability of Oregovomab When Added to Niraparib. | At week 7
  Humoral immune response measured by HAMA at week 7 relative to baseline.

OTHER OUTCOMES:
Progression-Free Survival (PFS) | Baseline up to two years
  Defined as date of first dose of study treatment to the date of event defined as the first documented progression as per RECIST v1.1
Overall Survival (OS) | Baseline up to two years
  Defined as the portion of subjects who survive for 24 months after first dose.
Overall Response Rate (ORR) | Week 12 to Week 24
  Overall Response Rate (ORR) to alternate next-line therapy-initiated post Week 12 measured at Week 24 relative to their Week 12 assessment ((new baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Gupta, MD, FRCPC, Study Director — CanariaBio Inc.
Locations (3):
- United States (3):
  - Duke Cancer Center, Durham, North Carolina
  - Stephenson Cancer Center- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No